CLINICAL TRIAL: NCT01489787
Title: A Phase I-II Study to Evaluate, in Patients Operated for a Hepatic Resection of Colorectal Liver Metastases, a High Intensity Focused Ultrasound (HIFU) Procedure: Feasibility, Safety and Accuracy.
Brief Title: Study to Evaluate a High Intensity Focused Ultrasound (HIFU) Procedure in Patient With Liver Metastases
Acronym: HIFU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government); Cancéropôle Lyon Auvergne Rhône-Alpes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU; ET2009-068 (Other: Sponsor number)
Record Dates: First submitted 2011-11-24; First posted 2011-12-12 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2017-01

CONDITIONS: Neoplasm Metastasis
Keywords: Surgery; Ultrasonic therapy; Liver
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase I : HIFU (Experimental)
  Interventions: Procedure: HIFU
- Phase IIa : HIFU (Experimental)
  Interventions: Procedure: HIFU
- Phase IIb : HIFU (Experimental)
  Interventions: Procedure: HIFU

INTERVENTIONS:
Procedure: HIFU — The shootings will concern the healthy liver to remove, distant to the important vascular structures and metastases. Two HIFU shootings will be made on each patient:
  * One hurt on the surface starting from the Glisson capsule and extending to subjacent hepatic parenchyma.
  * One hurt at given depth, at least 10 mm deeper than the hurt done on the surface NB: The shooting depth will determined for each patient at the beginning of the operation, considering preoperative exams (scans, etc.), size and location of the liver part to be resected and physical structure of the patient.
  Arms: Phase I : HIFU
Procedure: HIFU — The shootings will concern healthy liver to be resected, distant (step 1) then close (step 2) to the important vascular structures of the liver. Several shootings HIFU will be made on each patient (ideally 4 hurts, minimum 2 hurts)
  Arms: Phase IIa : HIFU
Procedure: HIFU — Shootings will concern small metastases (≤ 20 mm) and peri lesional healthy liver. They will be juxtaposed on multiple plans in order to generate a large hurt containing the metastasis targeted and guaranteeing a sufficient safety margin in healthy liver.
  Several metastases can be treated in the same patient
  Arms: Phase IIb : HIFU

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of High Intensity Focused Ultrasound (HIFU) patients undergoing hepatectomy for colorectal liver metastases. This is a phase I/II study.

DETAILED DESCRIPTION:
Justification and interest of the study:

Colorectal liver metastases (CLM) are a major public health issue (16 000 deaths each year in France). To date, complete resection of CLM offers the only potential curative approach. However, only a minority of patients (10 to 20%) is candidates. 5-year survival rates after liver resection are ranged from 20 to 35%. Consequently, alternative locally targeted therapies (radiofrequency, cryotherapy, laser, microwave) have been developed and evaluated. Their use presents many limitations: invasive procedures requiring the intraparenchymal introduction of a probe, impossibility of an accurate monitoring in real-time, small size destruction, time-consuming, high recurrence rate. The development of a non-invasive and more accurate technique combined to surgery is required.

High Intensity Focused Ultrasound (HIFU) is a new approach, which enables to generate irreversible cell death through coagulative necrosis in a few seconds. There's no cooling effect of the perfusion because of the shortness of the phenomenon.

The surgical team of the Centre Leon Berard, in collaboration with the INSERM U556 one, has undertaken a research program on CLM treatment by HIFU. A new and very powerful device, without the previously named limitations, has been developed. Preclinical studies have revealed the interest, the feasibility and the safety of this process. These results enable considering preceding the program with an early clinical study.

Experimental design:

Prospective, monocentric phase I/II study evaluating a surgical medical device (SMD).

HIFU SMD will be evaluated in clinical conditions, in patients undergoing hepatectomy for colorectal liver metastases. Several HIFU "shootings" (the number will be function of the advancement of the study) will be performed on the liver witch will be resected

Objectives and main assessment criteria:

1. st part: Phase I - on the healthy liver to remove. Feasibility 1, Safety 2, Tolerance 3. Success = 1 Ability to perform shootings, supplementary duration of intervention < 30 minutes; 2 Asepsis, absence of lesion of nearly tissues; 3 Preservation of hemodynamic and respiratory constants.
2. nd part: Phase IIa - on the healthy liver to remove, distant then close to the vascular structures of the liver.

   Ability of targeting shootings. Success = distance from the epicentre of the HIFU lesion to the mark previously positioned in the liver ≤ 5mm.
3. rd part: Phase IIb - on metastases to remove. Ability, by summation of HIFU lesions, to generate " macro-lesions " including a metastasis and insuring a sufficient safety margin in the healthy tissue.

Success = macro-lesion generated in negative margins.

Number of patients:

1. st part: The inclusion from 2 to 6 patients is required. The next step (phase II) will depend on:

   * 1st analysis after 2 patients:

     * If < 2 failures: continuation,
     * If 2 failures: cessation of the study.
   * 2nd analysis after 6 patients:

     * If < 3 failures: continuation (phase II),
     * If ≥ 3 failures: cessation.
2. nd part: Three patients will be successively included in each of the 2 landings (appendix 1):

   * If no failure: continuation (2nd landing / Phase IIb),
   * If ≤ 2 failures: + 3 patients,
   * If > 2 failures on 6 patients: cessation,
   * If ≤ 2 failures on 6 patients: continuation (2nd landing / phase IIb),
   * If 3 failures: cessation.
3. rd part:

   * p0 = 0.70 = upper limit of the success rate resulting in the inefficacy of HIFU multi-shootings.
   * p1 = 0.90 = lower limit of the success rate resulting in the efficacy of HIFU shootings.

With a 5% risk of type I error and a 80% power, 28 metastases have to be targeted by HIFU in order to conclude in one-sided situation. Taking into account that an average of 1.5 metastases will be targeted in each patient, 20 patients will be enrolled. 24 observed successes will allow concluding in the reject of H0 to accept H1.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more patient,
* Affected of hepatic metastasis of a colorectal cancer,
* Who must undergo a hepatectomy by laparotomy with the aim of the resection of hepatic metastasis,
* ECOG performance status (PS) = 1,
* Mandatory affiliation to a health security insurance,
* Written informed consent.

Exclusion Criteria:

* Having already undergone a major hepatic surgery (more than three segments) or biliary major (context of major iterative hepatic surgery),
* Having already undergone a major abdominal surgery with the exception of a colorectal surgery for the treatment of its primitive tumor (the surgery of the gall-bladder by laparoscopy for the deadline upper to 6 months do not constitute a criterion of not inclusion),
* Unable to be followed during the duration of the study,
* Pregnant or breast-feeding woman (a pregnancy test must be negative at the time of the inclusion in the study for the women in age to procreate; a method of reliable contraception must be used during the duration of the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2010-03 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
First step: Ability to shoot and supplementary duration of intervention, to use the medical device following requested asepsis procedures and no evidence of hurt on peripheral tissues and to keep vital signs stable | At the end of surgery (realized about 1 week after enrollment)
Phase IIa - First step: accuracy of shootings on a precise area | At the end of surgery (realized about 1 week after enrollment)
  both the distance between the hurt epicentre generated by hifu and a mark. These sizes will be measured in mm during anatomopathological exam.
Phase IIb: possibility of ≤ 15 shootings, safety margin ≥ 5 mm in healthy liver. | At the end of surgery (realized about 1 week after enrollment)
Phase IIa - Second step: accuracy of shootings on a zone to be spared | At the end of surgery (realized about 1 week after enrollment)
  between the hurt limit and a vessel border previously marked. These sizes will be measured in mm during anatomopathological exam.

SECONDARY OUTCOMES:
Phase I: adjust the probe position to different liver segments and patient physical structure. | At the end of surgery (realized about 1 week after enrollment)
  The aim is to be free to generate a HIFU hurt in at least 80 % of the total liver volume
Phase I: Possibility to set a stationary mark, at given depth, echographically detectable | At the end of surgery (realized about 1 week after enrollment)
Phase I: Possibility to spot echographically a previously Patent Blue or Methylene blue marked vessel | At the end of surgery (realized about 1 week after enrollment)
Phase I: Mean duration to achieve each step expressed in minutes(initialization, conditioning, targeting, shooting) | At the end of surgery (realized about 1 week after enrollment)
Phase I: description of outline during perioperative echography | At the end of surgery (realized about 1 week after enrollment)
  diameters, depth, volume
Phase I: description of limits during anatomopathological analysis | At the end of surgery (realized about 1 week after enrollment)
  diameters, depth, volume
Phase I: distance between the mark / marked vessel and the hurt limits during anatomopathological analysis | At the end of surgery (realized about 1 week after enrollment)
  Precise measure given in mm by the anatomopathologist
Phase II: safety of the device | At the end of surgery (realized about 1 week after enrollment)
  no evidence of hurt on peripheral tissues (Glisson capsule on the opposite side of the HIFU shootings entrance area, retro-peritoneal, retro-hepatic tissues and diaphragm
Phase II: assessment of vital signs during shooting phase | At the end of surgery (realized about 1 week after enrollment)
  hemodynamic, respiratory, body temperature
Phase IIa: correlation between hurt perioperative echographic and postoperative macroscopic, measures | At the end of surgery (realized about 1 week after enrollment)
  hurt dimensions comparison (diameters, depth, volume, etc. - in mm), blind-measured, with echography in a first time and in a second time, right after the resection, in anatomopathology

CONTACTS AND LOCATIONS:
Overall Officials: Michel RIVOIRE, Principal Investigator — Centre Léon Bérard, LYON, FRANCE
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Manfredi S, Lepage C, Hatem C, Coatmeur O, Faivre J, Bouvier AM. Epidemiology and management of liver metastases from colorectal cancer. Ann Surg. 2006 Aug;244(2):254-9. doi: 10.1097/01.sla.0000217629.94941.cf. PMID 16858188
- [Background] Bismuth H, Adam R, Levi F, Farabos C, Waechter F, Castaing D, Majno P, Engerran L. Resection of nonresectable liver metastases from colorectal cancer after neoadjuvant chemotherapy. Ann Surg. 1996 Oct;224(4):509-20; discussion 520-2. doi: 10.1097/00000658-199610000-00009. PMID 8857855
- [Background] Mulier S, Ni Y, Jamart J, Ruers T, Marchal G, Michel L. Local recurrence after hepatic radiofrequency coagulation: multivariate meta-analysis and review of contributing factors. Ann Surg. 2005 Aug;242(2):158-71. doi: 10.1097/01.sla.0000171032.99149.fe. PMID 16041205
- [Background] Rivoire M, De Cian F, Meeus P, Negrier S, Sebban H, Kaemmerlen P. Combination of neoadjuvant chemotherapy with cryotherapy and surgical resection for the treatment of unresectable liver metastases from colorectal carcinoma. Cancer. 2002 Dec 1;95(11):2283-92. doi: 10.1002/cncr.10973. PMID 12436433
- [Background] Antoniou A, Lovegrove RE, Tilney HS, Heriot AG, John TG, Rees M, Tekkis PP, Welsh FK. Meta-analysis of clinical outcome after first and second liver resection for colorectal metastases. Surgery. 2007 Jan;141(1):9-18. doi: 10.1016/j.surg.2006.07.045. Epub 2006 Nov 17. PMID 17188163
- [Background] Pawlik TM, Schulick RD, Choti MA. Expanding criteria for resectability of colorectal liver metastases. Oncologist. 2008 Jan;13(1):51-64. doi: 10.1634/theoncologist.2007-0142. PMID 18245012
- [Background] Garcea G, Lloyd TD, Aylott C, Maddern G, Berry DP. The emergent role of focal liver ablation techniques in the treatment of primary and secondary liver tumours. Eur J Cancer. 2003 Oct;39(15):2150-64. doi: 10.1016/s0959-8049(03)00553-7. PMID 14522372
- [Background] Seifert JK, Morris DL. Indicators of recurrence following cryotherapy for hepatic metastases from colorectal cancer. Br J Surg. 1999 Feb;86(2):234-40. doi: 10.1046/j.1365-2168.1999.00995.x. PMID 10100794
- [Background] Coleman DJ, Lizzi FL, Driller J, Rosado AL, Burgess SE, Torpey JH, Smith ME, Silverman RH, Yablonski ME, Chang S, et al. Therapeutic ultrasound in the treatment of glaucoma. II. Clinical applications. Ophthalmology. 1985 Mar;92(3):347-53. doi: 10.1016/s0161-6420(85)34028-9. PMID 3991122
- [Background] Valtot F, Kopel J, Petit E, Moulin F, Haut J. [Treatment of refractory glaucoma with high density focused ultrasonics]. J Fr Ophtalmol. 1995;18(1):3-12. French. PMID 7738293
- [Background] Chapelon JY, Margonari J, Vernier F, Gorry F, Ecochard R, Gelet A. In vivo effects of high-intensity ultrasound on prostatic adenocarcinoma Dunning R3327. Cancer Res. 1992 Nov 15;52(22):6353-7. PMID 1423282
- [Background] Poissonnier L, Chapelon JY, Rouviere O, Curiel L, Bouvier R, Martin X, Dubernard JM, Gelet A. Control of prostate cancer by transrectal HIFU in 227 patients. Eur Urol. 2007 Feb;51(2):381-7. doi: 10.1016/j.eururo.2006.04.012. Epub 2006 May 2. PMID 16857310
- [Background] Kinsey AM, Diederich CJ, Rieke V, Nau WH, Pauly KB, Bouley D, Sommer G. Transurethral ultrasound applicators with dynamic multi-sector control for prostate thermal therapy: in vivo evaluation under MR guidance. Med Phys. 2008 May;35(5):2081-93. doi: 10.1118/1.2900131. PMID 18561684
- [Background] Madersbacher S, Pedevilla M, Vingers L, Susani M, Marberger M. Effect of high-intensity focused ultrasound on human prostate cancer in vivo. Cancer Res. 1995 Aug 1;55(15):3346-51. PMID 7542168
- [Background] Vallancien G, Harouni M, Guillonneau B, Veillon B, Bougaran J. Ablation of superficial bladder tumors with focused extracorporeal pyrotherapy. Urology. 1996 Feb;47(2):204-7. doi: 10.1016/S0090-4295(99)80417-8. PMID 8607235
- [Background] Wu F, Wang ZB, Cao YD, Zhu XQ, Zhu H, Chen WZ, Zou JZ. "Wide local ablation" of localized breast cancer using high intensity focused ultrasound. J Surg Oncol. 2007 Aug 1;96(2):130-6. doi: 10.1002/jso.20769. PMID 17443737
- [Background] Melodelima D, Prat F, Fritsch J, Theillere Y, Cathignol D. Treatment of esophageal tumors using high intensity intraluminal ultrasound: first clinical results. J Transl Med. 2008 Jun 5;6:28. doi: 10.1186/1479-5876-6-28. PMID 18533990
- [Background] Wu F, Wang ZB, Chen WZ, Zhu H, Bai J, Zou JZ, Li KQ, Jin CB, Xie FL, Su HB. Extracorporeal high intensity focused ultrasound ablation in the treatment of patients with large hepatocellular carcinoma. Ann Surg Oncol. 2004 Dec;11(12):1061-9. doi: 10.1245/ASO.2004.02.026. Epub 2004 Nov 15. PMID 15545506
- [Background] Vaezy S, Fujimoto VY, Walker C, Martin RW, Chi EY, Crum LA. Treatment of uterine fibroid tumors in a nude mouse model using high-intensity focused ultrasound. Am J Obstet Gynecol. 2000 Jul;183(1):6-11. doi: 10.1067/mob.2000.105347. PMID 10920300
- [Background] Marquet F, Pernot M, Aubry JF, Montaldo G, Marsac L, Tanter M, Fink M. Non-invasive transcranial ultrasound therapy based on a 3D CT scan: protocol validation and in vitro results. Phys Med Biol. 2009 May 7;54(9):2597-613. doi: 10.1088/0031-9155/54/9/001. Epub 2009 Apr 8. PMID 19351986
- [Background] Uchida T, Ohkusa H, Nagata Y, Hyodo T, Satoh T, Irie A. Treatment of localized prostate cancer using high-intensity focused ultrasound. BJU Int. 2006 Jan;97(1):56-61. doi: 10.1111/j.1464-410X.2006.05864.x. PMID 16336329
- [Background] Melodelima D, N'Djin WA, Parmentier H, Chesnais S, Rivoire M, Chapelon JY. Thermal ablation by high-intensity-focused ultrasound using a toroid transducer increases the coagulated volume. Results of animal experiments. Ultrasound Med Biol. 2009 Mar;35(3):425-35. doi: 10.1016/j.ultrasmedbio.2008.09.020. Epub 2008 Dec 10. PMID 19081666
- [Background] Parmentier H, Melodelima D, N'Djin A, Chesnais S, Chapelon JY, Rivoire M. High-intensity focused ultrasound ablation for the treatment of colorectal liver metastases during an open procedure: study on the pig. Ann Surg. 2009 Jan;249(1):129-36. doi: 10.1097/SLA.0b013e31818c70b6. PMID 19106688
- [Background] N'Djin WA, Melodelima D, Parmentier H, Chesnais S, Rivoire M, Chapelon JY. Utility of a tumor-mimic model for the evaluation of the accuracy of HIFU treatments. results of in vitro experiments in the liver. Ultrasound Med Biol. 2008 Dec;34(12):1934-43. doi: 10.1016/j.ultrasmedbio.2008.04.012. Epub 2008 Jul 14. PMID 18621469
- [Background] Lee YJ, Wesley RA. Statistical contributions to phase II trials in cancer: interpretation, analysis and design. Semin Oncol. 1981 Dec;8(4):403-16. No abstract available. PMID 7323812
- [Background] A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001 Mar 30;20(6):859-66. doi: 10.1002/sim.721. PMID 11252008
- [Derived] Dupre A, Rivoire M, Metzger S, Cropet C, Vincenot J, Peyrat P, Chen Y, Perol D, Melodelima D. Intra-operative High-Intensity Focused Ultrasound in Patients With Colorectal Liver Metastases: A Prospective Ablate-and-Resect Study. Ultrasound Med Biol. 2023 Aug;49(8):1845-1851. doi: 10.1016/j.ultrasmedbio.2023.04.010. Epub 2023 May 31. PMID 37268553
- [Derived] Dupre A, Melodelima D, Perol D, Chen Y, Vincenot J, Chapelon JY, Rivoire M. First clinical experience of intra-operative high intensity focused ultrasound in patients with colorectal liver metastases: a phase I-IIa study. PLoS One. 2015 Feb 26;10(2):e0118212. doi: 10.1371/journal.pone.0118212. eCollection 2015. PMID 25719540